CLINICAL TRIAL: NCT04269824
Title: The Longitudinal Evaluation of Norms and Networks Study: A Cluster Randomized Controlled Trial to Promote Exclusive Toilet Use in Tamil Nadu, India
Brief Title: The Norms and Networks Sanitation Study in India in Tamil Nadu, India
Acronym: LENNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 833854
Record Dates: First submitted 2020-02-05; First posted 2020-02-17 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Behavior, Social; Norms, Social
Keywords: Sanitation; Norms; Toilet Use; Toilet Ownership
MeSH Terms: conditions — Social Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Residents of the peri-urban ward randomized to this group will receive the norm and network-centric intervention package that includes individual, household, group and community-level interventions. No hardware will be provided. Behavior change components will focus on shifting empirical expectations of improved sanitation behaviors in their wards as well as building capacity to achieve toilet construction and behavioral goals.
  Interventions: Behavioral: Behavioral intervention package
- Control Group (No Intervention): Residents of these wards will not receive any intervention. They may be exposed to other WASH interventions promoted by the government and/or other parties independent of this study.

INTERVENTIONS:
Behavioral: Behavioral intervention package — Community mobilization and commitment events
  * Update factual beliefs
  * Establish public commitment
  * Update empirical expectations about toilet use
  Audio announcements - Disseminate norms-related messages regarding toilet use and ownership
  Group level
  - Facilitated sex-segregated group meetings to share information and action knowledge through increased social connections
  Network-level social media messages - Transmit norms-related messages, and testimonials of adopters through influential social network members
  Household-level Counseling visits
  * Update empirical expectations of improved sanitation behaviors in their community
  * Motivate improved sanitation practices
  * Build capacity to achieve exclusive toilet use
  Stickers/decals
  - Signal adoption of promoted behaviors to community members
  Individual-level
  * Update empirical expectations of improved behaviors among similar others
  * Set goals, track progress and maintain improved behavior
  Arms: Intervention Group

SUMMARY:
The objective of this research is to evaluate the impact of a multi-level behavior change intervention designed to promote toilet construction, exclusive toilet use and maintenance in peri-urban communities of Tamil Nadu. The intervention leverages two years of formative research and reflects a norms and network-centric approach that will employ dynamic information dissemination to signal others' sanitation practices while also addressing other barriers to the adoption of improved sanitation practices. The study will determine whether those who received the interventions had significant improvements in toilet usage compared to those who did not. Qualitative research will help assess exposure and reactions to the intervention in these communities.

DETAILED DESCRIPTION:
The objective of this research is to evaluate the impact of a multi-level behavior change intervention designed to promote toilet construction, exclusive toilet use and maintenance in peri-urban communities of Tamil Nadu. The intervention leverages two years of formative research and reflects a norms and network-centric approach that will employ dynamic information dissemination to signal others' sanitation practices while also addressing other barriers to the adoption of improved sanitation practices. The study will determine whether those who received the interventions had significant improvements in toilet usage compared to those who did not.

For this cluster-randomized trial, communities will be engaged in two rounds of surveys to assess toilet ownership, toilet usage practices of their family members and include additional questions about beliefs, norms and other factors influencing toilet use. Investigators will also conduct a process evaluation to monitor change from baseline to endline and identify successful pathways of or bottle-necks to the adoption of improved sanitation behaviors. These indicators will include fidelity indicators to assess the quality of intervention delivery, level of community participation, behavioral antecedents, contextual changes in community and household conditions that may facilitate improved behavioral adoption and/or outcomes (e.g., exclusive toilet use). They will also conduct qualitative research using observations and semi-structured interviews with respondents and stakeholders to assess exposure and reactions to the intervention. They will also assess spillover in the control wards using mixed-method assessment tools.

ELIGIBILITY:
Inclusion Criteria:

* Site: Peri-urban wards with 60% or less toilet coverage from selected town panchayats in Tamil Nadu.

Participants

* Randomly selected residents of eligible wards above 18 years of age.
* All households in the intervention wards will receive the LENNS intervention.

Exclusion Criteria:

* Site: Slum wards as they will not be representative of our population of interest.
* Wards that were included in the piloting of the intervention package.
* Wards enrolled in any water, sanitation or hygiene intervention other than the national program, Swachh Bharat Mission (SBM)

Participants:

* Persons who were reported or deemed cognitively unable to participate in the study and respond to the surveys will be excluded
* Household members who confirm that they will not reside continuously at that address in the upcoming year
* Specific household members who do not reside at that residency continuously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22700 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Change in exclusive toilet usage rate | Measured 12 months after intervention
  Exclusive toilet use is measured using self reported use of toilet every time for defecation in the past 2 days. It will be assessed via household survey conducted by trained enumerators and respondents.

SECONDARY OUTCOMES:
Change in Empirical expectations (beliefs of what other's do) regarding toilet ownership, use and maintenance | Measured 12 months after intervention
  Empirical expectation of toilet ownership, use and maintenance refers to individual's self reported belief of the prevalence of other's toilet ownership, use and maintenance respectively in their own community. It will be assessed via household survey using pre-tested indicators.
Change in the proportion of households with improved sanitation facilities | Measured 12 months after intervention
  An improved sanitation facility is defined as one that hygienically separates human excreta from human contact (WHO/UNICEF JMP 2019). It will be assessed through a household survey and direct observations of the sanitation facility by the surveyors.
Change in normative expectations (beliefs of what other think you should do) regarding toilet ownership, use and maintenance | Measured 12 months after intervention
  Normative expectation of toilet ownership, use and maintenance refers to individual's belief of the prevalence of whether the toilet ownership, use and maintenance is approved by others in their community. It will be assessed via household survey using pre-tested indicators.
Change in the usable toilet facilities rates | Measured 12 months after intervention
  Usable or functional toilet facility will be defined according using WHO/UNICEF JMP 2019 definitions and ascertained during direct observations of toilet facilities during household surveys.

OTHER OUTCOMES:
Change in diarrhea prevalence in children under 5 years | Measured 12 months after intervention
  Diarrhea is defined as 3+ loose or watery stools in 24 hours or 1+ stools with blood in 24 hours. This outcome will be assessed via a household survey conducted between the trained enumerators and participants.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Bicchieri, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Swasti, Bangalore, India

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD for the surveyed respondents will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be available after the completion of the RCT and will be open access.
Access Criteria: Open access with an application form
URL: https://normsandbehavior.sas.upenn.edu/lenns/

REFERENCES:
- [Derived] Ashraf S, Bicchieri C, Delea MG, Das U, Chauhan K, Kuang J, Shpenev A, Thulin E. Norms and Social Network-Centric Behavior Change Intervention (Nam Nalavazhvu) for Improved Toilet Usage in Peri-Urban Communities of Tamil Nadu: Protocol for a Cluster-Randomized Controlled Trial. JMIR Res Protoc. 2021 May 3;10(5):e24407. doi: 10.2196/24407. PMID 33938805

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-09-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT04269824/SAP_000.pdf